CLINICAL TRIAL: NCT00625872
Title: Neuromuscular Changes In Small For Gestational Age (SGA) Children During Somatropin Therapy - A Prospective Randomized, Controlled, Open-Label Multicenter Trial
Brief Title: Neuromuscular Changes In Small For Gestational Age Children During Somatropin Therapy
Acronym: SGA-POWER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study terminated on 19-Jan-2011 due to insufficient recruitment of patients. No safety reasons contributed to the termination of the study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6281283
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-01

CONDITIONS: Growth Hormone Therapy; Infant, Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): Somatropin for 12 months
  Interventions: Drug: Somatropin
- Control Group (Other): In the first 6 months no intervention, afterwards Somatropin for 12 months
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Patients will be randomized at baseline in a 1:1 ratio into treatment group or control group. After six months the control group will undergo GH therapy with a higher dose of 0.067 mg/kg/day, too. All patients are treated with growth hormone for 12 months.
  Arms: Treatment Group
Drug: Somatropin — Patients will be randomized at baseline in a 1:1 ratio into treatment group or control group. After six months the control group will undergo GH therapy with a higher dose of 0.067 mg/kg/day, too. All patients are treated with growth hormone for 12 months.
  Arms: Control Group

SUMMARY:
The planned study focuses on the effect of a one year Somatropin treatment (0.035 mg/kg/d or 0.067 mg/kg/d) in short children born SGA on neuromuscular function and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pubertal boys between 6 and 10 years of age or girls between 6 and 9 years of age.
* Birth length- and/or birth weight-SDS adjusted to gestational age < -2.0 (Voigt et al. 2002, Voigt et al. 2006 or Lawrence et al. 1989).
* Current height-SDS < -2.5 (Brandt/Reinken 1992) and parental adjusted height-SDS below -1 (Hermanussen and Cole 2003).
* Growth velocity SDS < 0 during the last year before inclusion (Brandt/Reinken 1988).

Exclusion Criteria:

* Severe SGA (birth weight or length < -4 SD) and clinically relevant dysmorphic features.
* Severe pre-maturity (GA < 32 weeks of gestation).
* Severe perinatal complications like asphyxia, sepsis, necrotizing enterocolitis (NEC), respiratory distress syndrome, if associated with long-term sequelae (like short bowel syndrome, bronchopulmonary dysplasia (BPD), cerebral palsy etc).
* Inability to perform one- or two leg jumps from a standing position.
* Prior GH treatment.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Germany (10):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Datteln
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Kiel
  - Pfizer Investigational Site, München

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281283&StudyName=Neuromuscular%20Changes%20In%20Small%20For%20Gestational%20Age%20Children%20During%20Somatropin%20Therapy

RESULTS

PARTICIPANT FLOW:
Groups:
- Somatropin: Somatropin 0.035 milligram/kilogram/day (mg/kg/day) was administered subcutaneously (s.c) according to exact body weight specific calculation for 12 months. Dose adjustments were made at 6 month intervals.
- Control Arm: No treatment for initial 6 months in control group, after 6 months, somatropin 0.067 mg/kg/day administered s.c. according to exact body weight specific calculation for 12 months.
Period: Overall Study
Arm/Group | Somatropin | Control Arm
Started | 12 | 11
Treated | 12 | 10
Completed | 8 | 5
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Does not meet inclusion criteria | 1 | 0
Not completed — Terminated by sponsor | 2 | 5
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Somatropin: Somatropin 0.035 mg/kg/day was administered s.c according to exact body weight specific calculation for 12 months. Dose adjustments were made at 6 month intervals.
- Total: Total of all reporting groups
Arm/Group | Somatropin | Control Arm | Total
Number analyzed (Participants) | 12 | 11 | 23
Age Continuous [Mean (Standard Deviation); unit: Years] | 6.6 (1.0) | 7.6 (1.4) | 7.1 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Jump Power Standard Deviation Score (PJP-SDS; Two-leg-jump) in Full Analysis Set (FAS) Population at Month 6
Description: Peak jump power (PJP) was defined as the peak of the calculated power (force multiplied by velocity). It was measured by Leonardo Jumping Platform during two-leg jump. The participant performs 3 jumps and the highest peak (PJP) of the 3 recordings was selected for further calculations. The SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline and Month 6
Population: FAS population included participants who received at least 1 dose of study medication and had at least one post baseline efficacy assessment. Number of participants analyzed (N) signifies participants evaluable for the measure.
Measure: Least Squares Mean (Standard Error); unit: Watt/kilogram (W/kg)
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 4 | 8
Watt/kilogram (W/kg) | -0.15 (1.01) [upper limit 3.07] | 0.28 (0.51) [upper limit 1.91]
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Analysis of covariance (ANCOVA) method was used to calculate p-value with treatment, baseline value, study duration and site as covariates; Test type: Superiority or Other; p = 0.7232, ANCOVA — The statistical test was 2-sided and performed at the 5 percent significance level; Least squares (LS) mean difference = -0.43, 95% CI 2-sided [-3.93 to 3.08], Standard Error of Mean 1.10

2. Primary Outcome: Change From Baseline in Peak Jump Power Standard Deviation Score (PJP-SDS; Two-leg-jump) in Per Protocol (PP) Population at Month 6
Description: PJP was defined as the peak of the calculated power (force multiplied by velocity). It was measured by Leonardo Jumping Platform during two-leg jump. The participant performs 3 jumps and the highest peak (PJP) of the 3 recordings was selected for further calculations. The SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline and Month 6
Population: PP population included participants who received the study medication for at least 22 weeks. Number of participants analyzed (N) signifies participants evaluable for the measure.
Measure: Least Squares Mean (Standard Error); unit: W/kg
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 2 | 6
W/kg | -1.02 (0.43) | 0.59 (0.27)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; ANCOVA method was used to calculate p-value with treatment, baseline value, study duration and site as covariates; Test type: Superiority or Other; p = 0.1941, ANCOVA — The statistical test was 2-sided and performed at the 5 percent significance level; LS Mean difference = -1.61, 95% CI 2-sided [-8.04 to 4.82], Standard Error of Mean 0.51

3. Primary Outcome: Change From Baseline in Peak Jump Force Standard Deviation Score (PJF-SDS; Two-leg-jump) in Full Analysis Set (FAS) Population at Month 6
Description: PJF was defined as the maximum of force of the ascending part of the jump which the participant performed as a counter-movement jump with freely moving arms and as high as possible with the head and chest. It was measured by Leonardo Jumping Platform during two-leg jump. The SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Newtons
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 4 | 8
Newtons | -0.70 (0.62) [upper limit 1.29] | -0.55 (0.29) [upper limit 0.38]

4. Secondary Outcome: Change From Baseline in Intellectual Performance of Children Using Kaufmann-Assessment Battery for Children (K-ABC) Test Global Scales at Month 6
Description: K-ABC was assessed in children between 2.5-12.5 years. Comprised of 16 subtests; 10 mental processing (intelligence) and 6 achievement subtests. Achievement subtests: expressive vocabulary, faces&places, arithmetic, riddles, reading/decoding, reading/comprehension. Sixteen subtests were weighted accordingly to form 5 global scales: sequential processing, simultaneous processing, achievement, non-verbal and mental processing composite. Scores were rated as upper extreme [greater than (>) 131], above average (116-130), average (85-115), below average (70-84), lower extreme [less than (<) 69].
Time Frame: Baseline and Month 6
Population: FAS population included participants who received at least 1 dose of study medication and had at least one post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 11 | 11
Units on a scale
  Baseline (Sequential Processing) | 25.7 (8.35) | 28.5 (8.33)
  Change at Month 6 (Sequential Processing) | 2.6 (5.82) | -1.9 (4.15)
  Baseline (Simultaneous Processing) | 45.7 (7.20) | 49.8 (12.74)
  Change at Month 6 (Simultaneous Processing) | -0.1 (4.53) | 1.5 (4.30)
  Baseline (Achievement) | 300.7 (66.83) | 341.8 (76.88)
  Change at Month 6 (Achievement) | 32.1 (48.79) | 16.7 (27.52)
  Baseline (Nonverbal) | 46.2 (8.65) | 49.8 (13.21)
  Change at Month 6 (Nonverbal) | -1.4 (3.78) | 0.0 (5.35)
  Baseline (Mental Processing Composite) | 70.0 (12.38) | 78.1 (19.95)
  Change at Month 6 (Mental Processing Composite) | 1.4 (6.39) | -0.9 (7.28)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; For K-ABC Test (Sequential Processing): Kruskal-Wallis Analysis of Variance (ANOVA) model was used to calculate p-value; Test type: Superiority or Other; p = 0.0532, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; For K-ABC Test (Simultaneous Processing): Kruskal-Wallis ANOVA model was used to calculate p-value; Test type: Superiority or Other; p = 0.3383, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level
Statistical Analysis 3: Comparison: Somatropin vs Control Arm; For K-ABC Test (Achievement): Kruskal-Wallis ANOVA model was used to calculate p-value; Test type: Superiority or Other; p = 0.6830, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level
Statistical Analysis 4: Comparison: Somatropin vs Control Arm; For K-ABC Test (Non-Verbal): Kruskal-Wallis ANOVA model was used to calculate p-value; Test type: Superiority or Other; p = 0.4935, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level
Statistical Analysis 5: Comparison: Somatropin vs Control Arm; For K-ABC Test (Mental Processing Composite): Kruskal-Wallis ANOVA model was used to calculate p-value; Test type: Superiority or Other; p = 0.3458, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level

5. Secondary Outcome: Change From Baseline in Intellectual Performance of Children Using Kaufmann-Assessment Battery for Children (K-ABC) Test Global Scales at Months 12 and 18
Description: as for outcome 4
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Intellectual Performance of Children Using Kinderversion Der Testbatterie Zur Aufmerksamkeitsprüfung für Kinder (KITAP) Test at Month 6
Description: The KITAP is a computer aided standardized neuro-cognitive development test which allows examination of a wide range of attention and executive functions such as shift of attention (Distractibility); simple reaction time (Alertness); "Sustained Attention", change of reaction (Flexibility); "Divided Attention", controlled reaction disposition (Go/No go) and "Vigilance". It has been designed appropriately for children between the age of 6 to 10 years to allow optimal motivation during testing and to increase validity of results.
Time Frame: Baseline and Month 6
Population: FAS population included participants who received at least 1 dose of study medication and had at least one post baseline efficacy assessment. Number of participants analyzed (N) signifies participants evaluable for the measure and 'n' signifies participants who received the study drug and evaluated at the time point for each group respectively.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 9 | 11
Seconds
  Baseline (Distractibility) | 554.3 (201.08) [300.0 to 978.0] | 514.5 (127.41) [321.0 to 709.0]
  Change at 6 Month (Distractibility) (n= 7, 10) | 5.6 (230.95) [-440.0 to 280.0] | -11.4 (139.52) [-223.0 to 216.0]
  Baseline (Alertness) | 433.9 (140.74) [250.0 to 626.0] | 384.6 (124.94) [245.0 to 573.0]
  Change at 6 Month (Alertness) (n= 8, 10) | -16.1 (80.85) [-150.0 to 119.0] | 4.0 (107.42) [-122.0 to 196.0]
  Baseline (Flexibility) | 1350.0 (470.50) [728.0 to 2001.0] | 1313.0 (477.19) [759.0 to 2140.0]
  Change at 6 Month (Flexibility) (n= 8, 10) | -192.0 (492.73) [-704.0 to 875.0] | -211.0 (589.41) [-1034.0 to 1189.0]
  Baseline (Go/No Go) | 539.8 (106.73) [362.0 to 691.0] | 514.9 (91.95) [399.0 to 730.0]
  Change at 6 Month (Go/No Go) (n= 8, 9) | 35.6 (113.38) [-95.0 to 208.0] | -50.2 (69.90) [-133.0 to 45.0]
  Baseline (Vigilance) | 822.2 (200.65) [569.0 to 1195.0] | 693.4 (118.01) [525.0 to 967.0]
  Change at 6 Month (Vigilance) (n= 7, 10) | -146.0 (278.60) [-627.0 to 265.0] | -31.2 (107.62) [-194.0 to 172.0]
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; For KITAP Test (Distractibility): Kruskal-Wallis ANOVA model was used to calculate p-value; Test type: Superiority or Other; p = 0.6256, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; For KITAP Test (Alertness): Kruskal-Wallis ANOVA model was used to calculate p-value; Test type: Superiority or Other; p = 0.8590, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level
Statistical Analysis 3: Comparison: Somatropin vs Control Arm; For KITAP Test (Flexibility): Kruskal-Wallis ANOVA model was used to calculate p-value; Test type: Superiority or Other; p = 1.0000, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level
Statistical Analysis 4: Comparison: Somatropin vs Control Arm; For KITAP Test (Go/No Go): Kruskal-Wallis ANOVA model was used to calculate p-value; Test type: Superiority or Other; p = 0.1234, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level
Statistical Analysis 5: Comparison: Somatropin vs Control Arm; For KITAP Test (Vigilance): Kruskal-Wallis ANOVA model was used to calculate p-value; Test type: Superiority or Other; p = 0.3291, Kruskal-Wallis — The statistical test was 2-sided and performed at the 5 percent significance level

7. Secondary Outcome: Change From Baseline in Intellectual Performance of Children Using Kinderversion Der Testbatterie Zur Aufmerksamkeitsprüfung für Kinder (KITAP) Test at Months 12 and 18
Description: as for outcome 6
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Intellectual Performance of Children Using Non-verbal Learning Test (NVLT) at Month 6
Description: NVLT was assessed for visual memorization that was difficult to verbalize. Test recorded instability index, T-scores[sum of differences of correct {C} - incorrect {IC} "Yes" answers(1);sum of C "Yes" answers(2);sum of IC "Yes" answers(3);sum of differences of C-IC "Yes" answers with high associative items{ 87%-95%}(4);sum of differences of C-IC "Yes" answers with low associative items{ 54%-64%}(5); difference between difference values for high and low associative items(6)].Scores were rated as below average(<40), average(40-60), above average(>60) and working time ranging between 9-12 minutes.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 9 | 11
Units on a scale
  Baseline (Instability Index) | 0.3 (0.15) | 0.2 (0.21)
  Change at Month 6 (Instability Index) | -0.1 (0.11) | -0.1 (0.20)
  Baseline (Working Time) | 227.0 (44.27) | 218.3 (76.89)
  Change at Month 6 (Working Time) | 10.6 (92.95) | -11.1 (34.86)
  Baseline [T-scores (1)] | 39.9 (13.60) | 43.9 (16.53)
  Change at Month 6 [T-scores (1)] | 4.4 (11.64) | 6.7 (12.12)
  Baseline [T-scores (2)] | 41.6 (12.97) | 46.8 (14.40)
  Change at Month 6 [T-scores (2)] | 5.0 (10.72) | -0.6 (5.50)
  Baseline [T-scores (3)] | 45.9 (14.89) | 48.1 (18.20)
  Change at Month 6 [T-scores (3)] | 1.5 (5.15) | 8.3 (12.24)
  Baseline [T-scores (4)] | 39.3 (16.97) | 46.4 (16.03)
  Change at Month 6 [T-scores (4)] | 5.6 (15.53) | 1.4 (11.75)
  Baseline [T-scores (5)] | 43.3 (11.12) | 43.6 (15.13)
  Change at Month 6 [T-scores (5)] | 2.6 (9.83) | 7.7 (12.59)
  Baseline [T-scores (6)] | 44.9 (15.83) | 52.9 (19.96)
  Change at Month 6 [T-scores (6)] | 0.9 (16.55) | -7.4 (14.88)
  Baseline [Age-corrected T-scores (1)] | 33.4 (12.18) | 38.6 (13.43)
  Change at Month 6 [Age-corrected T-scores (1)] | 6.0 (10.21) | 5.2 (11.26)
  Baseline [Age-corrected T-scores (2)] | 51.3 (7.55) | 54.5 (8.10)
  Change at Month 6 [Age-corrected T-scores (2)] | 3.1 (5.59) | -0.1 (3.38)
  Baseline [Age-corrected T-scores (3)] | 40.0 (13.86) | 41.1 (16.38)
  Change at Month 6 [Age-corrected T-scores (3)] | 0.6 (4.47) | 7.8 (12.13)
  Baseline [Age-corrected T-scores (4)] | 37.4 (17.01) | 45.0 (15.21)
  Change at Month 6 [Age-corrected T-scores (4)] | 6.3 (14.57) | 4.1 (10.63)
  Baseline [Age-corrected T-scores (5)] | 35.0 (11.88) | 37.3 (13.48)
  Change at Month 6 [Age-corrected T-scores (5)] | 3.3 (10.73) | 6.9 (12.57)
  Baseline [Age-corrected T-scores (6)] | 50.0 (16.49) | 55.5 (16.64)
  Change at Month 6 [Age-corrected T-scores (6)] | 1.5 (19.06) | -4.1 (13.77)

9. Secondary Outcome: Change From Baseline in Intellectual Performance of Children Using Non-verbal Learning Test (NVLT) at Months 12 and 18
Description: as for outcome 8
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Intellectual Performance of Children Using Child Behavior Checklist 4-18 Years (CBCL 4-18) at Months 6, 12 and 18
Description: CBCL was standardized for children ages 4 to 18 years and measured child internalizing and externalizing behaviors and total problems. The 4-18 years' checklist contains 140 questions and responses were recorded on a Likert scale: 0 = Not True, 1 = Somewhat or Sometimes True, 2 = Very True or Often True. The range of possible values was 0-280 (0=good to 280=worst).
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Peak Jump Power Standard Deviation Score (PJP-SDS; One-leg-jump) at Months 6, 12 and 18
Description: PJP was defined as the peak of the calculated power (force multiplied by velocity). It was measured by Leonardo Jumping Platform during one leg jump. The participant performs 3 jumps and the highest peak (PJP) of the 3 recordings was selected for further calculations. The SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 6 , Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Peak Jump Force Standard Deviation Score (PJF-SDS; One-leg-jump) at Months 6, 12 and 18
Description: PJF was defined as the maximum of force of the ascending part of the jump which the participant performed as a counter-movement jump with freely moving arms and as high as possible with the head and chest. It was measured by Leonardo Jumping Platform during one leg jump. The SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Maximum Jump Velocity (Vmax; One-leg-jump) at Months 6, 12 and 18
Description: Vmax was measured by Leonardo Jumping Platform during one leg jump.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in Five-chair Rising Test- Peak Jump Power (PJP) at Month 6
Description: The Chair rising test is a performance test (total power output) to measure neuromuscular function of complex movement in standing up. Test allows diagnostics of movement deficits using Leonardo jump plate. Five stand up test: five repetitions of rising from a chair on jump plate as quickly as possible with arms crossed over the chest (time to perform the tasks, maximal PJP, maximal velocity and maximal PJF). PJP is defined as the peak of the calculated power (force multiplied by velocity).
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilowatt (kW)
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 9 | 9
kilowatt (kW)
  Baseline | 0.1 (0.07) | 0.1 (0.05)
  Change at Month 6 | 0.0 (0.07) | 0.0 (0.05)

15. Secondary Outcome: Change From Baseline in Five-chair Rising Test-Peak Jump Power (PJP) at Months 12 and 18
Description: as for outcome 14
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: kW
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in Five-chair Rising Test-Peak Jump Force (PJF) at Month 6
Description: The Chair rising test is a performance test (total power output) to measure neuromuscular function of complex movement in standing up. Test allows diagnostics of movement deficits using Leonardo jump plate. Five stand up test: five repetitions of rising from a chair on jump plate as quickly as possible with arms crossed over the chest (time to perform the tasks, maximal PJP, maximal velocity and maximal PJF). PJF is the maximum force of the ascending part of the jump which the participant performed as a counter-movement jump with freely moving arms as high as possible with the head and chest.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilonewton (kN)
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 9 | 9
kilonewton (kN)
  Baseline | 0.4 (0.11) | 0.4 (0.19)
  Change at Month 6 | -0.0 (0.23) | 0.0 (0.20)

17. Secondary Outcome: Change From Baseline in Five-chair Rising Test-Peak Jump Force (PJF) at Months 12 and 18
Description: as for outcome 16
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: kN
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change From Baseline in Five-chair Rising Test-Maximum Jump Velocity (Vmax) at Month 6
Description: The Chair rising test is a performance test (total power output) to measure neuromuscular function of complex movement in standing up. Test allows diagnostics of movement deficits using Leonardo jump plate. Five stand up test: five repetitions of rising from a chair on jump plate as quickly as possible with arms crossed over the chest (time to perform the tasks, maximal PJP, maximal velocity and maximal PJF). Vmax is defined as the maximum jump velocity.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 9 | 9
m/s
  Baseline | 0.7 (0.22) | 0.6 (0.16)
  Change at Month 6 | 0.2 (0.29) | 0.0 (0.18)

19. Secondary Outcome: Change From Baseline in Five-chair Rising Test-Maximum Jump Velocity (Vmax) at Months 12 and 18
Description: as for outcome 18
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in Five-chair Rising Test (Time to Perform the Tasks) at Month 6
Description: Chair rising test is performance test (total power output) to measure neuromuscular function of complex movement in standing up. Test allows diagnostics of movement deficits using Leonardo jump plate. Five stand up test: 5 repetitions of rising from a chair on jump plate as quickly as possible with arms crossed over chest (time to perform tasks, maximal PJP, maximal velocity and maximal PJF). Time to perform task includes: Average (avg) rise time which is avg time to perform 1 rise, avg time per test is the avg time to perform 1 test (rise and sitting down) and total time to perform 5 tests.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 9 | 9
seconds
  Baseline (Average rise time) | 1.2 (0.90) | 0.7 (0.31)
  Change at Month 6 (Average rise time) | -0.5 (1.15) | 0.1 (0.27)
  Baseline (Average time per test) | 2.0 (0.70) | 2.3 (0.60)
  Change at Month 6 (Average time per test) | -0.2 (0.54) | -0.1 (0.87)
  Baseline (Total time to perform 5 tests) | 9.6 (3.91) | 10.8 (2.24)
  Change at Month 6 (Total time to perform 5 tests) | 0.1 (3.04) | 2.0 (8.48)

21. Secondary Outcome: Change From Baseline in Five-chair Rising Test (Time to Perform the Tasks) at Months 12 and 18
Description: as for outcome 20
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Baseline in One-chair Rising Test-Peak Jump Power (PJP) at Months 6, 12 and 18
Description: The Chair rising test is a performance test (total power output) to measure neuromuscular function of complex movement to stand up. Test allows diagnostics of movement deficits using Leonardo jump plate. One stand up test: rising from a chair on the jump plate as quickly as possible with arms crossed over the chest (analysis of time, PJP, PJF and time of fastest rising). PJP is defined as the peak of the calculated power (force multiplied by velocity).
Time Frame: Baseline, Month 6 , Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: kW
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change From Baseline in One-chair Rising Test-Peak Jump Force (PJF) at Months 6, 12 and 18
Description: The Chair rising test is a performance test (total power output) to measure neuromuscular function of complex movement to stand up. Test allows diagnostics of movement deficits using Leonardo jump plate. One stand up test: rising from a chair on the jump plate as quickly as possible with arms crossed over the chest (analysis of time, PJP, PJF and time of fastest rising). PJF is the maximum force of the ascending part of the jump which the participant performed as a counter-movement jump with freely moving arms as high as possible with the head and chest.
Time Frame: Baseline, Month 6 , Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: kN
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Change From Baseline in One-chair Rising Test (Time to Perform the Tasks) at Months 6, 12 and 18
Description: The Chair rising test is a performance test (total power output) to measure neuromuscular function of complex movement to stand up. Test allows diagnostics of movement deficits using Leonardo jump plate. One stand up test: rising from a chair on the jump plate as quickly as possible with arms crossed over the chest (analysis of time, PJP, PJF and time of fastest rising).
Time Frame: Baseline, Month 6 , Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Change From Baseline in Maximal Isometric Grip Force-Standard Deviation Score (MIGF-SDS) at Month 6
Description: MIGF was assessed using standard adjustable Jamar dynamometer. MIGF (in Newtons) was calculated by multiplying the dynamometer reading (in kilograms) by a factor of 9.81. The SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 9 | 11
kg | 1.28 (1.69) | 1.13 (1.64)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; ANCOVA method was used to calculate p-value with treatment, baseline value, study duration and site as covariates; Test type: Superiority or Other; p = 0.9560, ANCOVA — The statistical test was 2-sided and performed at the 5 percent significance level; LS Mean difference = 0.14, 95% CI 2-sided [-5.71 to 6.00], Standard Error of Mean 2.54

26. Secondary Outcome: Change From Baseline in Maximal Isometric Grip Force-Standard Deviation Score (MIGF-SDS) at Months 12 and 18
Description: as for outcome 25
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

27. Other Pre Specified Outcome: Change From Baseline in Bone Density Using Peripheral Quantitative Computed Tomography (pqCT) at 6 or 12 or 18 Months
Description: Bone Mineral Density (BMD) was measured by pqCT. The Z-score measures the distance of the measured BMD value from the appropriate normal age matched population mean value in units of standard deviation of this population. More negative scores indicate less BMD compared to age matched population and more positive scores indicate higher BMD compared to age matched population.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

28. Other Pre Specified Outcome: Change From Baseline in Bone Structure Using Peripheral Quantitative Computed Tomography (pqCT) at 6 or 12 or 18 Months
Description: Bone structure was measured by pqCT.Parameters included:total area,cortical area,marrow area,cortical thickness,cortical density of the radius,bone strength,cross-sectional muscle and fat area,total bone density,bone mineral count,trabecular BMD,bone cross-sectional area.Baseline and post-baseline SDS values transformed to age and sex specific z-score([Ln(test result/M)]/S);Ln=natural logarithm;M=age-/height- and sex-specific mean value;S=age-/height- and sex-specific coefficient of variation).Positive values are above the average for participant's age and sex;negative values are below.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

29. Other Pre Specified Outcome: Change From Baseline in Bone Stability Using Peripheral Quantitative Computed Tomography (pqCT) at 6 or 12 or 18 Months
Description: Bone stability was measured by pqCT. Baseline and post-baseline SDS values transformed to age and sex specific z-score (Ln(test result/M)]/S); Ln=natural logarithm; M=age- (or height-) and sex-specific mean value; S=age-(or height-) and sex-specific coefficient of variation) then change from baseline is calculated. Positive values are above the average for participant's age and sex; negative values are below the average.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Mean Upper Arm Circumference
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Mean Thigh Circumference
Description: Thigh measurements were taken as a mean of 3 consecutive measurements at upper thigh about an inch down from the crotch line.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Mean Calf Circumference
Description: Calf measurements were taken as a mean of 3 consecutive measurements at largest part of calf muscle, usually about 4 inches down from below the knee.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Mean Height at Month 6
Description: Standing height was taken as a mean of 3 consecutive measurements using a wall mounted stadiometer.
Time Frame: Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 11 | 11
cm | 112.8 (5.13) | 115.0 (7.93)

34. Secondary Outcome: Mean Height at Months 12 and 18
Description: Standing height was taken as a mean of 3 consecutive measurements using a wall mounted stadiometer.
Time Frame: Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Mean Growth Velocity at Month 6
Description: Growth velocity measures the annual rate of increase in height.
Time Frame: Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 11 | 11
cm/year | 8.2 (1.93) | 4.6 (1.44)

36. Secondary Outcome: Mean Growth Velocity at Months 12 and 18
Description: Growth velocity measures the annual rate of increase in height.
Time Frame: Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Mean Height-Standard Deviation Score (SDS) at Month 6
Description: Standing height was taken as a mean of 3 consecutive measurements using a wall mounted stadiometer. The SDS indicates how similar the participant was to the reference population.
Time Frame: Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 11 | 11
cm | -3.1 (0.86) | -3.7 (0.77)

38. Secondary Outcome: Mean Height-Standard Deviation Score (SDS) at Months 12 and 18
Description: as for outcome 37
Time Frame: Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Mean Growth Velocity-Standard Deviation Score (SDS) at Month 6
Description: Growth velocity measures the annual rate of increase in height. The SDS indicates how similar the participant is to the reference population.
Time Frame: Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 11 | 11
cm/year | 3.4 (2.62) | -1.1 (1.43)

40. Secondary Outcome: Mean Growth Velocity-Standard Deviation Score (SDS) at Months 12 and 18
Time Frame: Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Change From Baseline in Height-Standard Deviation Score (SDS) at Month 6
Description: as for outcome 37
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 11 | 11
cm | 0.33 (0.21) | -0.22 (0.25)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; ANCOVA method was used to calculate p-value with treatment, baseline value, study duration and site as covariates; Test type: Superiority or Other; p = 0.1107, ANCOVA — The statistical test was 2-sided and performed at the 5 percent significance level; LS Mean difference = 0.55, 95% CI 2-sided [-0.15 to 1.25], Standard Error of Mean 0.31

42. Secondary Outcome: Change From Baseline in Height-Standard Deviation Score (SDS) at Months 12 and 18
Description: as for outcome 37
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Change From Baseline in Growth Velocity-Standard Deviation Score (SDS) at Month 6
Description: as for outcome 39
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 9 | 9
cm/year | 3.89 (1.02) | -0.77 (1.40)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; ANCOVA method was used to calculate p-value with treatment, baseline value, study duration and site as covariates; Test type: Superiority or Other; p = 0.0161, ANCOVA — The statistical test was 2-sided and performed at the 5 percent significance level; LS Mean difference = 4.67, 95% CI 2-sided [1.13 to 8.21], Standard Error of Mean 1.54

44. Secondary Outcome: Change From Baseline in Growth Velocity-Standard Deviation Score (SDS) at Months 12 and 18
Description: as for outcome 39
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

45. Primary Outcome: Change From Baseline in Peak Jump Force Standard Deviation Score (PJF-SDS; Two-leg-jump) in Per Protocol (PP) Population at Month 6
Description: as for outcome 3
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Newtons
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 2 | 6
Newtons | -0.83 (1.27) | -0.85 (0.73)

46. Primary Outcome: Change From Baseline in Maximum Jump Velocity (Vmax; Two-leg-jump) in Full Analysis Set (FAS) Population at Month 6
Description: Vmax was measured by Leonardo Jumping Platform during two-leg jump.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Meter/second (m/s)
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 10 | 11
Meter/second (m/s) | 0.01 (0.08) [upper limit 0.18] | 0.12 (0.09) [upper limit 0.32]

47. Primary Outcome: Change From Baseline in Maximum Jump Velocity (Vmax; Two-leg-jump) in Per Protocol (PP) Population at Month 6
Description: Vmax was measured by Leonardo Jumping Platform during two-leg jump.
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 5 | 9
m/s | 0.01 (0.05) | 0.25 (0.06)

48. Secondary Outcome: Sitting Height-Standard Deviation Score (SDS)
Description: Sitting height was measured using a stadiometer with a specialized chair. The SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Body Mass Index-Standard Deviation Score (BMI-SDS)
Description: The BMI was used to measure body fat based on height and weight. It was calculated by body weight (kg) divided by the height (m) squared. The SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

50. Secondary Outcome: Change From Baseline in Head Circumference at Months 6, 12 and 18
Description: The maximum head circumference (usually horizontal just above the eyebrow ridges), was measured from just above the glabella area to the area near the top of the occipital bone (opisthocranion).
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Change From Baseline in Head Circumference-Standard Deviation Score (SDS) at Months 6, 12 and 18
Description: The maximum head circumference (usually horizontal just above the eyebrow ridges), was measured from just above the glabella area to the area near the top of the occipital bone (opisthocranion). The SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 6, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Change From Baseline in Skinfold Thickness-Standard Deviation Score (SDS) at Month 6
Description: Triceps, supra-iliac and subscapular skinfolds were measured on the right side of the body to the nearest 0.1 mm with a Holtain skinfold caliper. The measurement was performed at the left side of the participant. Triceps skinfold thickness was measured halfway down the left upper arm, while the arm was hanging relaxed at the participant's side. Suprascapular skinfold was measured laterally just below the angle of the left scapula. Suprailiac skinfold was measured just above the iliac crest in the middle-axillary line. SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 11 | 11
Millimeter (mm)
  Change at Month 6 (Triceps SDS) | -0.41 (0.16) | -0.06 (0.18)
  Change at Month 6 (Subscapular SDS) | -0.30 (0.10) | -0.16 (0.13)
  Change at Month 6 (Suprailiac SDS) | -0.60 (0.07) | -0.33 (0.12)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Triceps SDS: ANCOVA method was used to calculate p-value with treatment, baseline value, study duration and site as covariates; Test type: Superiority or Other; p = 0.1870, ANCOVA — The statistical test was 2-sided and performed at the 5 percent significance level; LS Mean difference = -0.35, 95% CI 2-sided [-0.89 to 0.20], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Subscapular SDS: ANCOVA method was used to calculate p-value with treatment, baseline value, study duration and site as covariates; Test type: Superiority or Other; p = 0.3494, ANCOVA — The statistical test was 2-sided and performed at the 5 percent significance level; LS Mean difference = -0.15, 95% CI 2-sided [-0.49 to 0.19], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Somatropin vs Control Arm; Suprailiac SDS: ANCOVA method was used to calculate p-value with treatment, baseline value, study duration and site as covariates; Test type: Superiority or Other; p = 0.0458, ANCOVA — The statistical test was 2-sided and performed at the 5 percent significance level; LS Mean difference = -0.27, 95% CI 2-sided [-0.54 to -0.01], Standard Error of Mean 0.12

53. Secondary Outcome: Change From Baseline in Skinfold Thickness-Standard Deviation Score (SDS) at Months 12 and 18
Description: as for outcome 52
Time Frame: Baseline, Month 12 and Month 18
Population: Data were not analyzed as study was prematurely terminated due to insufficient number of participants.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Somatropin | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 10/12 | 7/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somatropin (N=12) | Control Arm (N=11)
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Lice infestation (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 0 | 1
Scarlet fever (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Lordosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Enuresis (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued, therefore not all data was powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.